## Imperial College London

Hammersmith Hospital, Du Cane Road, London W12 0HS P: 02033133000 W: <a href="https://www.imperial.nhs.uk">www.imperial.nhs.uk</a>

Email: keenan.saleh10@imperial.ac.uk

Study Protocol Number: IRAS 347921 Patient Identification Number for this trial:

Name of Person taking consent

(If different from Researcher)

## **Consent Form For Adults**

| Full Title of Project: Al-ECG Accessory Pathway Localisation Study | | |
|---|---|---|
| Naı | me of Principal Investigator: | Please initial box |
| 1. | I confirm that I have read and understand the participant information sheet version | |
| 2. | I understand that my participation is voluntary, and I am free to withdraw at any time, without giving any reason and without my legal rights nor treatment / healthcare being affected. | |
| 3. | I understand that sections of any of my medical notes may be looked at by responsible individuals from Imperial College Londo from NHS Trusts or from regulatory authorities where it is relevant my taking part in this research. | |
| 4. | I give/do not give (delete as applicable) consent for information collected about me to be used to support other research or in the development of a new test by an academic institution or commercompany in the future, including those outside of the United Kingdom (which Imperial has ensured will keep this information secure). | |
| 5. | I understand that data collected from me are a gift donated to Imperial College and that I will not personally benefit financially if this research leads to an invention and/or the successful development of a new test, medication treatment, product or service. | |
| 6. | I consent to take part in the AI-ECG Accessory Pathway Localisation study. | |
| 7. | I give / do not give (delete/mark as applicable) consent to being contacted about the possibility to take part in other research stud | ies. |
| | Name of Patient Date | Signature |

1 copy for participant; 1 copy for Principal Investigator 1 copy for hospital notes
To ensure confidence in the process and minimise risk of loss, all consent forms <u>must</u> be printed,
presented and stored in double sided format

Date

IRAS: 347921 Version 1 Date: 07/08/24



Signature